CLINICAL TRIAL: NCT06426875
Title: Effects Of Isometric Muscle Training On Shoulder Pain, Function And Performance In Bowlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01834 Sheeraz Ali Shaikh
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Shoulder Pain
Keywords: Isometric; Shoulder Pain; Bowlers; Performance
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Group 1 Experimental Group 2 Control
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects Of Isometric Muscle Training On Shoulder Pain, Function And Performance In Bowlers (Experimental): The Isometric Exercise Program which comprises targeted exercises for declining pain, improving function and performance, exercises were focused only on shoulder flexion, extension, abduction, adduction, internal rotation and external rotation. Exercises were performed via Thera Bands, free weights and resistance. Each repetition was of 10 to 15 seconds and 10 to 15 number of repetition total of three sets according to FITT formula. Under the supervision of a therapist, these exercises were performed three times each week. Every training session lasts 35 to 40 minutes, with a 5-minute warm-up and a 5-minute cool-down in between. Instruction in the correct form and technique was provided to participants throughout the intervention, and their development was closely evaluated to guarantee safety and effectiveness. Total duration of 35 to 40-minute session three sessions per week total four weeks of intervention, reading will be taken on baseline and after 2nd week and 4th week.
  Interventions: Diagnostic Test: Isometric Exercises
- Control Group (No Intervention): (control group) in this group participants will receive Traditional Physical therapy

INTERVENTIONS:
Diagnostic Test: Isometric Exercises — Isometric External Rotation (Perform isometric external rotation exercises with a resistance band to strengthen the rotator cuff.) Hold each contraction for 10-15 seconds. Isometric Internal Rotation (Hold each contraction for 10-15 seconds) Isometric Abduction (Supraspinatus). ( each contraction for 10 -15 sec) 10 repetition 3 sets Isometric Adduction (Subscapularis) Overhead Isometric Holds (Hold each contraction for 15-20 seconds) Isometric Shoulder External Rotation Against Resistance: (Hold each contraction for 15-20 seconds) Isometric Shoulder Press (Hold each contraction for 15-20 seconds) 15 to 20 repetitions 4 sets Total duration of 30 to 35 minute session three sessions per week total four weeks of intervention, reading will be taken on baseline and after 2nd week and 4th week
  Arms: Effects Of Isometric Muscle Training On Shoulder Pain, Function And Performance In Bowlers

SUMMARY:
Goal of this clinical trial is to determine whether Isometric muscle training decrease pain improve function and enhance performance.

Does Isometric exercise improve pain function and performance in bowlers? Researcher will compare the Isometric muscle training with Traditional therapy to examine that isometric exercise work on pain function and performance.

Participants will receive isometric exercises for three days in week and will be followed up after two weeks total four weeks of trial(experimental group).

Participants will receive traditional physical therapy treatment three days of week and followed up after two weeks total four weeks of trail (contril group)

DETAILED DESCRIPTION:
This research is critical for addressing a common health concern and providing evidence-based recommendations for a potentially effective and accessible intervention that can significantly enhance the quality of life and performance of individuals dealing with shoulder pain. Thesis will benefit the bowlers by increasing their performance by enhancing accuracy, speed and consistency and over all shoulder health. Because shoulder discomfort is so common and has such a detrimental influence on everyday activities and performance, research on how isometric muscle training affects shoulder pain, function, and performance is crucial. In a variety of settings, isometric training has demonstrated promise in enhancing musculoskeletal function and pain management; however, its precise influence on shoulder-related problems is yet unknown.

ELIGIBILITY:
Inclusion Criteria:

* Active Male Bowlers
* Age 18 - 30
* Pain that affects performance. Any level of pain that significantly affects a bowler's performance, accuracy, or consistency.
* Pain with psychological impact. Pain that causes emotional distress, anxiety, or frustration.
* Rotator Cuff pain.
* Weekly 6 to 8 hour training

Exclusion Criteria:

* Other than bowlers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Disability of Arm Hand and Shoulder (DASH) | 4th weeks
  The DASH questionnaire consists of 30 questions concerning upper limb function and symptoms. Patients figure out their ability to carry out each activity or the degree of their symptoms on a scale from 1 (no difficulty or no symptoms) to 5 (unable to perform the activity or vigorous symptoms). The results are then transformed into a standardized score, ranging from 0 to 100, with higher scores indicating more disabilities

SECONDARY OUTCOMES:
Manual Muscle Testing | 4th week
  It is used to assess weakness and also useful in identifying actual weakness from imbalance or inadequate endurance. It may be referred to as motor testing, muscular strength grading, manual muscle testing, or any other synonym
Visual Analogue Scale VAS | 4th week
  A VAS consists of a line, usually 10 cm long, with language anchors at each end, similar to an NRS (e.g., "no pain" on the far left and "the most intense pain imaginable" on the far right)
Bowling Speed Test | 4th week
  Bowling speed test: A bowling speed app is a mobile application made to measure and analyze the speed of a thrown cricket ball
Bowling Accuracy Test | 4th week
  (Cones, Target Set, Wicket to Wicket Bowling, and Video Analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Riafat Mehmood, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Elite Cricket Academy Shahbaz sharif sports complex, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Not sharing